CLINICAL TRIAL: NCT02934386
Title: Validation of the WBPS - Wrist Blood Pressure System A Prospective, Method Comparison, Proof of Concept Study
Brief Title: WBPS A Prospective, Method Comparison, Proof of Concept Study
Acronym: WBPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CSEM Centre Suisse d'Electronique et de Microtechnique SA - Recherche et Developpement (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: WBPS
Record Dates: First submitted 2016-10-13; First posted 2016-10-17 (Estimated); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- WinMedical WinPack device (Experimental): 50 volunteers undergoing experimental protocol according to IEEE 1708:2014 standard
  Interventions: Device: WinMedical WinPack device

INTERVENTIONS:
Device: WinMedical WinPack device

SUMMARY:
The study will evaluate the accuracy of BP measurements by a new algorithm to be embedded to the existing CE-marked WinPack device, compared to two reference devices (one oscillometric and one volume-clamp device), in healthy subjects and patients undergoing a standardized physical-activity hypertensive protocol.

DETAILED DESCRIPTION:
Current standard for patient monitoring in acute care such as intensive care units (ICU), operating rooms (OR) or emergency rooms (ER) is the use of expensive, bulky and uncomfortable monitors.

Unfortunately, once discharged from the acute care setting and transferred to a general division for example (low acuity), patients are left with manual measurements of vital signs every 4 to 6 hours, depending on the available resources in nursing. Furthermore, these measurements reflect only the results of the time the measurement is taken (spot check). The combination of manual spot checks and lack of innovative medical technology in 60% of hospital care settings (all non-ICUs and non-OR) represents an important limitation to patient follow-up, with its associated risks and costs.

In particular, when referring to the monitoring of blood pressure (BP), current monitoring practice relies on the use of occlusive pneumatic cuffs inflated around the arm. Based on oscillometric technique, occlusive cuffs not only are uncomfortable, but they provide only intermittent measurements, with the inability to provide a full view of the BP regulation landscape. Therefore, un-detected hypertensive events can be omitted, putting the patient at risk.

The continuous, comfortable and portable measurement of BP in low acuity hospital departments is a major unsolved problem of modern healthcare systems with regards to patient monitoring and safety.

Winmedical (device manufacturer) commercializes a wearable multi-parametric modular medical system, WinPack, to deliver continuous real-time monitoring and recording of vital signs, such as electrocardiography (ECG), respiration rate, BP, blood oxygen saturation, body temperature, and posture, in low-acuity departments to increase the overall clinical performance. A new algorithm to process the raw physiological signals acquired by the WinPack to provide more accurate and more continuous BP measurement is now to be tested.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Informed Consent
* Compliant and able to protocol manoeuvres

Exclusion Criteria:

* Blood pressure difference between to arms >15mmHg
* Current or history of tobacco smoking (for the last 5 years, > 5 cigarettes per day),
* Current alcohol or drug abuse (>4 units per day),
* Unstable cardiac condition (myocardial infarction < 1 week, pulmonary embolism, ventricular arrhythmia, decompensated heart failure)
* Severe anaemia (haemoglobin <100g/l)
* Oxygen therapy
* Lesion or deficiency on left hand, preventing to perform handgrip exercises
* Lesion or deficiency on both legs, preventing to perform leg extension exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-10; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Assessment of the accuracy of a novel algorithm to extract BP estimates from data acquired by the WinPack system, when compared to gold-standard BP devices, with respect to limits of agreement as stated by the IEEE 1708:2014 standard | 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Cyril Pellaton, Dr, Principal Investigator — HNE - Hôpital Neuchâtelois, Site de Pourtalès
Locations (1):
- HNE - Hôpital Neuchâtelois, Site de Pourtalès, Neuchâtel, Switzerland

IPD SHARING:
Plan to Share IPD: No